CLINICAL TRIAL: NCT01331239
Title: A Proof of Concept, Open-label, Forced Titration, Multi-center Study to Assess the Safety/Tolerability and Efficacy of 10-weeks Treatment of LCI699 in Patients With Cushing's Disease
Brief Title: Safety and Efficacy of LCI699 in Cushing's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCI699C2201; 2010-022403-22 (EudraCT Number)
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cushings Disease; Cushing Disease
Keywords: Cushing Disease; osilodrostat; LCI699; Pituitary Gland; Adrenocorticotropic Hormone
MeSH Terms: conditions — Adrenocortical Hyperfunction; Pituitary ACTH Hypersecretion; Pituitary Diseases | interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part l: Core cohort (Experimental): Participants took an ascending dose of LCI699 (osilodrostat) from 2mg bid or 5 mg bid, up to 30 mg bid and participated in Part I of this study. 4 patients in this cohort moved to Part II of the study
  Interventions: Drug: LCI699
- Part II Core: Expansion cohort (Experimental): Participants took an ascending dose from 2mg bid or 5 mg bid, up to 30 mg bid and participated in the Part II Core Expansion of this study. These patients were all newly enrolled into the phase II part of the study
  Interventions: Drug: LCI699
- Part II Core: Follow-up cohort (Experimental): Participants took an ascending dose from 2mg bid or 5 mg bid, up to 30 mg bid and participated in the Part II Core Follow-up of this study. These patients were patients who transferred from Part I Core phase of the study
  Interventions: Drug: LCI699

INTERVENTIONS:
Drug: LCI699 — Osilodrostat 1 mg and 5 mg capsules, was prepared by Novartis and supplied to the Investigator. The capsule formulation of osilodrostat was later changed to tablets and this change was implemented in the study with Protocol amendment 6. Osilodrostat was open labeled 1 mg, 5 mg, 10 mg and 20 mg tablets.
  Other Names: osilodrastat

SUMMARY:
This exploratory study is a proof of concept study to determine whether LCI699 can safely reduce the level of urinary free cortisol in patients with Cushing's disease.

In addition, this study evaluated the long term efficacy and safety of LCI699 including an additional 12 week of treatment followed by a 12 month long term optional extension.

A second extension provided patients who were clinically benefitting from LCI699 an opportunity to continue to have access to the drug until LCI699 was commercially available and reimbursed or through the availability of a local access program.

DETAILED DESCRIPTION:
The Primary objective of this study was to assess the effect of 10-week treatment osilodrostat on 24 hour urine free cortisol (UFC) in patients with Cushing's disease.

The study consisted of a screening period of up to 60 days (to allow an adequate washout period for any medications that modified cortisol levels), a 10-14-day baseline period, a 10-week sequential dose escalation treatment period and a 14-day washout period followed by a Study Completion evaluation approximately 14 days after the last drug administration. Twelve patients were recruited and completed Part l of the study.

Eligible patients were dosed at 2 mg b.i.d for the first two weeks, the dose could then be increased every two weeks as necessary (to doses of 5, 10, 20 and 50 mg b.i.d). If at anytime, the subject's UFC was < Upper Limit of Normal (ULN), dose escalation was halted and the subject remained on the current, efficacious dose through Week 10, with continued monitoring of UFC responses every 2 weeks to allow continued dose adjustments if necessary. If at any time the subject experienced side effects which were either intolerable or met dose adjustment criteria, the prescribed dose was adjusted.

The primary endpoint (UFC ≤ ULN or ≥50% decrease at Day 70) was achieved by all patients. Subsequently, in order to confirm these observations, protocol was amended (Protocol amendment 4) and new patients were enrolled and investigated for a longer treatment period.

Following Protocol amendment 4, the study design was modified to include patients in Part II of the study for evaluating the long-term efficacy and safety of osilodrostat treatment for 22 weeks. Nineteen patients (15 who were treated in the expansion cohort in Part ll and 4 who participated in Part l) with Cushing's disease were enrolled as part of the Expansion cohort in Part II of the study. The 12 patients who had entered the study in Part I, were allowed to re-enter the study as the Core proof of concept (PoC) Follow-up cohort. At Day 70 ± 2 days (Week 10), all patients (both patients entering for the first time and those reentering the study) entered the 12-week assessment period. At Day 154, patients completed the End of Treatment-Core visit.

On Day 154 (Week 22), patients had the option to enter the 12-month extension phase (long-term extension 1). On Day 490, patients who continued in the study had the option to enter a second long term extension phase (extension-2) at the Investigator's discretion, provided they did not meet any of the study discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Cushing's Disease (persistent or recurrent) as evidenced by increased 24-hour urine free cortisol (UFC), normal or increased morning plasma Adrenocorticotropic Hormone (ACTH), and pituitary origin of excess ACTH.
* Patients with de novo Cushing's disease can be included only if they are not considered candidate for surgery

Exclusion Criteria:

* Patients treated with mitotane 6 months prior to Visit 1
* Patients with compression of the optic chiasm
* Patients with a known inherited syndrome as the cause for hormone over secretion
* Patients with Cushing's syndrome due to ectopic ACTH secretion or adrenal Cushing's syndrome
* Patients with pseudo-Cushing's syndrome
* Patients who are not biochemically euthyroid
* Diabetic patients with poorly controlled diabetes (HbA1c >9%)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after completion of dosing.
* Patients who have received pituitary irradiation within five years prior to Visit 1.
* Patients with risk factors for QTc prolongation or Torsade de Pointes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03-23 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (4):
  - Northwestern University Endo, Metabolism and Molecular, Chicago, Illinois
  - Massachusetts General Hospital Neuroendocrine Unit, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University SC, Portland, Oregon
- France (2):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Paris
- Italy (2):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Napoli
- Japan (2):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Chiba

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fleseriu M, Pivonello R, Lacroix A, Biller BMK, Feelders R, Gadelha M, Bertherat J, Belaya Z, Piacentini A, Pedroncelli AM, Newell-Price J. Osilodrostat dose impact on efficacy/safety in Cushing's disease: large, pooled analysis of LINC 2, 3, and 4. Eur J Endocrinol. 2025 Oct 30;193(5):606-617. doi: 10.1093/ejendo/lvaf207. PMID 41052284
- [Derived] Bertagna X, Pivonello R, Fleseriu M, Zhang Y, Robinson P, Taylor A, Watson CE, Maldonado M, Hamrahian AH, Boscaro M, Biller BM. LCI699, a potent 11beta-hydroxylase inhibitor, normalizes urinary cortisol in patients with Cushing's disease: results from a multicenter, proof-of-concept study. J Clin Endocrinol Metab. 2014 Apr;99(4):1375-83. doi: 10.1210/jc.2013-2117. Epub 2013 Dec 11. PMID 24423285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 were enrolled in the study: 12 in Part l and 19 in Part ll Core. Four of the participants in the Part II Core were previously enrolled in the Part I Core.
  That is, 4 participants who were included in Part 1 as well as in Part 2, re-enrolled in the study in part 2 (i.e., they completed the informed consent process again in Part 2, and were considered re-enrolled, after originally enrolling in part 1).
Pre-assignment Details: For overall study: 27 patients were planned; For Part l of the study, 12 - 15 patients were planned to be enrolled. For Part ll Core 19 patients were planned to be enrolled.
Groups:
- Part l: Core Cohort: Participants took an ascending dose of LCI699 (osilodrostat) from 2mg bid or 5 mg bid, up to 30 mg bid and participated in Part l of this study. 4 patients in this cohort moved to Part II of the study
- Part II Core: Expansion Cohort: Participants took an ascending dose from 2mg bid or 5 mg bid, up to 30 mg bid and participated in the Part ll Core Expansion of this study. These patients were all newly enrolled into the phase ll part of the study.
- Part ll Core: Follow-up Cohort: Participants took an ascending dose from 2mg bid or 5 mg bid, up to 30 mg bid and participated in the Part ll Core Follow-up of this study. These patients were patients who transferred from Part l Core phase of the study.
Period: Part I: Core Study
Arm/Group | Part l: Core Cohort | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Started | 12 | 0 | 0
Completed | 12 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part II: Core Study
Arm/Group | Part l: Core Cohort | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Started | 0 | 15 | 4
Completed | 0 | 7 | 3
Not Completed | 0 | 8 | 1
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Subj's cond. no longer require treatment | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Administrative problems | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Part l: Core cohort: safety analysis set (SAS): All subjects that received at least one dose of study drug.
  Part 2: Expansion cohort: Full Analysis Set (FAS): All patients in Follow-up cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part l: Core Cohort | Part II Core: Expansion Cohort | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Customized [Number; unit: Participants]
  <65 years | 12 | 15 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 12 | 11 | 23
  Black or African American | 0 | 3 | 3
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders to LCI699 Based on the Change in Mean Urinary Free Cortisol (UFC) From Baseline to Week 10
Description: A patient was considered to be a responder if his/her mean UFC level from the three 24-hour urine samples collected at Week 10 was ≤ Upper Limit of Normal (ULN), as defined by the local laboratories, or represented a ≥50% decrease from baseline. Patients who discontinued for a disease or treatment related reason (e.g. death, adverse event, clinical disease progression etc.), or whose mean Week 10 24-hour UFC levels were higher than the normal limit and experienced <50% decrease in UFC were classified as non-responders.
Time Frame: 10 weeks
Population: Primary Analysis Set: All patients with evaluable UFC data (at least two 24 hour measurements for both baseline and Week 10) were included in the primary efficacy analysis set. Of the 12 patients enrolled to this arm, 9 of the 12 patients met this criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Part l: Core Cohort
Number analyzed (Participants) | 9
Percentage of participants | 100.0

2. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of Hypothalamic-Pituitary-Adrenal (HPA)-Axis: 11- Deoxycorticosterone (Overall)
Description: Change in Deoxycorticosterone over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: Safety Analysis Set (SAS): All patients in the Core proof of concept (PoC) follow-up cohort who received at least one dose of study treatment after reentering the study and all patients in the Expansion cohort who received at least one dose of study treatment after Protocol amendment 04.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
pmol/L
  BL: 11-Deoxycorticosterone: number analyzed (Participants) | 12 | 4
  BL: 11-Deoxycorticosterone | 292.8 (371.54) | 188.0 (105.21)
  WK 22: 11-Deoxycorticosterone: number analyzed (Participants) | 10 | 4
  WK 22: 11-Deoxycorticosterone | 6957.8 (9627.77) | 3670.0 (2734.34)
  WK 70: 11-Deoxycorticosterone: number analyzed (Participants) | 7 | 4
  WK 70: 11-Deoxycorticosterone | 2523.1 (1597.39) | 1743.0 (1048.22)
  LOV: 11-Deoxycorticosterone: number analyzed (Participants) | 12 | 4
  LOV: 11-Deoxycorticosterone | 1640.8 (2097.16) | 1822.3 (1452.72)

3. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: 11-Deoxycortisol (Overall)
Description: Change in Deoxycortisol over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: Safety Analysis Set (SAS): All patients in the Core PoC follow-up cohort who received at least one dose of study treatment after reentering the study and all patients in the Expansion cohort who received at least one dose of study treatment after Protocol amendment 04.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
nmol/L
  BL: 11-Deoxycortisol: number analyzed (Participants) | 14 | 4
  BL: 11-Deoxycortisol | 4.21 (4.648) | 5.48 (6.549)
  WK 22: 11-Deoxycortisol: number analyzed (Participants) | 12 | 4
  WK 22: 11-Deoxycortisol | 45.48 (44.880) | 54.75 (60.676)
  WK 70: 11-Deoxycortisol: number analyzed (Participants) | 9 | 4
  WK 70: 11-Deoxycortisol | 15.32 (13.463) | 9.03 (7.934)
  LOV: 11-Deoxycortisol: number analyzed (Participants) | 14 | 4
  LOV: 11-Deoxycortisol | 8.60 (18.910) | 11.83 (19.101)

4. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Aldosterone, Thyroxine, Free (T4)
Description: Change in aldosterone & thyroxine, free over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
pmol/L
  BL: Aldosterone: number analyzed (Participants) | 14 | 4
  BL: Aldosterone | 165.5 (255.07) | 127.0 (177.04)
  WK 22: Aldosterone: number analyzed (Participants) | 12 | 4
  WK 22: Aldosterone | -151.1 (290.53) | -64.5 (247.93)
  WK 70: Aldosterone: number analyzed (Participants) | 9 | 4
  WK 70: Aldosterone | -101.9 (153.82) | -120.0 (182.11)
  LOV: Aldosterone: number analyzed (Participants) | 14 | 4
  LOV: Aldosterone | -135.1 (258.36) | -99.5 (149.06)
  BL: Thyroxine, free: number analyzed (Participants) | 14 | 4
  BL: Thyroxine, free | 14.02 (3.233) | 18.40 (8.050)
  WK 22: Thyroxine, free: number analyzed (Participants) | 11 | 4
  WK 22: Thyroxine, free | -1.17 (3.254) | -3.63 (3.247)
  WK 70: Thyroxine, free: number analyzed (Participants) | 9 | 4
  WK 70: Thyroxine, free | 0.46 (2.355) | -3.78 (7.951)
  LOV: Thyroxine, free: number analyzed (Participants) | 14 | 4
  LOV: Thyroxine, free | 1.69 (3.281) | -2.33 (5.324)

5. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Estradiol (Female)
Description: Change in Estradiol in females over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: Safety Analysis Set (SAS): All patients in the Core PoC follow-up cohort who received at least one dose of study treatment after reentering the study and all patients in the Expansion cohort who received at least one dose of study treatment after Protocol amendment 04. This analysis was on the female patients only.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 11 | 3
pmol/L
  BL: Female Estradiol: number analyzed (Participants) | 10 | 3
  BL: Female Estradiol | 209.60 (282.423) | 307.23 (263.028)
  WK 22: Female Estradiol: number analyzed (Participants) | 8 | 3
  WK 22: Female Estradiol | -42.19 (223.444) | -24.63 (234.288)
  WK 70: Female Estradiol: number analyzed (Participants) | 6 | 3
  WK 70: Female Estradiol | 10.55 (187.443) | -141.00 (376.080)
  LOV: Female Estradiol: number analyzed (Participants) | 10 | 3
  LOV: Female Estradiol | -114.24 (305.334) | 666.93 (1108.794)

6. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Estradiol (Male)
Description: Change in Estradiol in males over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: Safety Analysis Set (SAS): All patients in the Core PoC follow-up cohort who received at least one dose of study treatment after reentering the study and all patients in the Expansion cohort who received at least one dose of study treatment after Protocol amendment 04. This analysis was on the male patients only.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 4 | 1
pmol/L
  BL: Male Estradiol | 55.00 (25.755) | 77.10 (NA) — NA: Standard Deviation (SD) could not be calculated as there was only 1 patient.
  WK 22: Male Estradiol | 35.00 (68.005) | 18.30 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 70: Male Estradiol: number analyzed (Participants) | 3 | 1
  WK 70: Male Estradiol | -1.00 (16.523) | 110.10 (NA) — NA: SD could not be calculated as there was only 1 patient.
  LOV: Male Estradiol | 2.50 (55.729) | -33.10 (NA) — NA: SD could not be calculated as there was only 1 patient.

7. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Follicle Stimulation Hormone (FSH) (Female)
Description: Change in FSH in females over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 11 | 3
U/L
  BL: Female FSH: number analyzed (Participants) | 10 | 3
  BL: Female FSH | 9.09 (13.277) | 2.43 (0.929)
  WK 22: Female FSH: number analyzed (Participants) | 7 | 3
  WK 22: Female FSH | 14.89 (28.673) | 2.90 (2.476)
  WK 70: Female FSH: number analyzed (Participants) | 6 | 3
  WK 70: Female FSH | 3.58 (14.021) | 3.20 (2.081)
  LOV: Female FSH: number analyzed (Participants) | 10 | 3
  LOV: Female FSH | 15.41 (23.613) | 3.70 (2.524)

8. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Follicle Stimulation Hormone (Male)
Description: Change in FSH in males over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 4 | 1
U/L
  BL: Male FSH | 5.88 (3.241) | 5.80 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 22: Male FSH | -1.20 (1.560) | -5.20 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 70: Male FSH: number analyzed (Participants) | 3 | 1
  WK 70: Male FSH | -1.80 (1.735) | -5.80 (NA) — NA: SD could not be calculated as there was only 1 patient.
  LOV: Male FSH | -1.38 (5.660) | -2.90 (NA) — NA: SD could not be calculated as there was only 1 patient.

9. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Renin, Insulin, Thyrotropin
Description: Change in Renin, Insulin & Thyrotropin over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
mU/L
  BL: Renin: number analyzed (Participants) | 14 | 4
  BL: Renin | 23.706 (18.0642) | 73.973 (102.338)
  WK 22: Renin: number analyzed (Participants) | 12 | 4
  WK 22: Renin | 45.899 (144.9575) | -16.838 (145.6609)
  WK 70: Renin: number analyzed (Participants) | 9 | 4
  WK 70: Renin | 70.051 (117.9931) | -55.638 (88.9155)
  LOV: Renin: number analyzed (Participants) | 14 | 4
  LOV: Renin | 24.209 (52.0438) | -43.718 (70.5958)
  BL: Insulin: number analyzed (Participants) | 14 | 4
  BL: Insulin | 25.61 (27.166) | 22.38 (7.071)
  WK 22: Insulin: number analyzed (Participants) | 12 | 4
  WK 22: Insulin | -10.63 (20.247) | -8.58 (4.456)
  WK 70: Insulin: number analyzed (Participants) | 9 | 4
  WK 70: Insulin | -8.69 (24.132) | -12.53 (8.772)
  LOV: Insulin: number analyzed (Participants) | 14 | 4
  LOV: Insulin | -8.11 (23.169) | -5.78 (11.771)
  BL: Thyrotropin: number analyzed (Participants) | 14 | 4
  BL: Thyrotropin | 0.659 (0.6827) | 0.815 (0.8364)
  WK 22: Thyrotropin: number analyzed (Participants) | 11 | 3
  WK 22: Thyrotropin | 1.445 (2.3295) | 0.280 (0.3118)
  WK 70: Thyrotropin: number analyzed (Participants) | 9 | 4
  WK 70: Thyrotropin | 2.387 (4.0991) | 0.395 (0.4674)
  LOV: Thyrotropin: number analyzed (Participants) | 14 | 4
  LOV: Thyrotropin | 1.244 (3.4627) | 0.885 (0.5994)

10. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Insulin-like Growth Factor-1
Description: Change in Insulin-like Growth Factor-1 over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
ug/L
  BL: Insulin-like Growth Factor-1: number analyzed (Participants) | 14 | 3
  BL: Insulin-like Growth Factor-1 | 157.56 (109.044) | 235.30 (110.249)
  WK 22: Insulin-like Growth Factor-1: number analyzed (Participants) | 12 | 3
  WK 22: Insulin-like Growth Factor-1 | -9.78 (67.387) | -35.20 (153.817)
  WK 70: Insulin-like Growth Factor-1: number analyzed (Participants) | 9 | 3
  WK 70: Insulin-like Growth Factor-1 | -41.23 (76.969) | -113.43 (86.529)
  LOV: Insulin-like Growth Factor-1: number analyzed (Participants) | 14 | 3
  LOV: Insulin-like Growth Factor-1 | -56.76 (105.936) | -46.07 (62.155)

11. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Luteinising Hormone (LH) (Female)
Description: Change in LH in females over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 11 | 3
U/L
  BL: Female LH: number analyzed (Participants) | 10 | 3
  BL: Female LH | 2.78 (2.220) | 1.00 (1.000)
  WK 22: Female LH: number analyzed (Participants) | 8 | 2
  WK 22: Female LH | 7.45 (17.051) | 4.40 (0.990)
  WK 70: Female LH: number analyzed (Participants) | 6 | 3
  WK 70: Female LH | 7.47 (15.267) | 2.63 (3.235)
  LOV: Female LH: number analyzed (Participants) | 10 | 3
  LOV: Female LH | 7.30 (10.885) | 3.37 (2.060)

12. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: LH (Male)
Description: Change in LH in males over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 4 | 1
U/L
  BL: Male LH | 2.48 (1.328) | 5.90 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 22: Male LH | 0.48 (1.081) | -5.70 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 70: Male LH: number analyzed (Participants) | 3 | 1
  WK 70: Male LH | -0.53 (1.021) | -5.90 (NA) — NA: SD could not be calculated as there was only 1 patient.
  LOV: Male LH | -0.05 (2.610) | -2.70 (NA) — NA: SD could not be calculated as there was only 1 patient.

13. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Testosterone (Female)
Description: Change in Testosterone in females over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 11 | 3
nmol/L
  BL: Female Testosterone: number analyzed (Participants) | 10 | 3
  BL: Female Testosterone | 1.18 (0.820) | 1.43 (0.404)
  WK 22: Female Testosterone: number analyzed (Participants) | 8 | 3
  WK 22: Female Testosterone | 1.85 (1.790) | 5.27 (5.353)
  WK 70: Female Testosterone: number analyzed (Participants) | 6 | 3
  WK 70: Female Testosterone | 0.53 (1.409) | 0.50 (1.400)
  LOV: Female Testosterone: number analyzed (Participants) | 10 | 3
  LOV: Female Testosterone | 0.25 (1.532) | 0.17 (1.266)

14. Secondary Outcome: Actual Change From Baseline (BL) in Steroid Hormones of HPA-axis: Testosterone (Male)
Description: Change in Testosterone in males over time.
Time Frame: baseline, Week 22, Week 70, Last observed value (LOV), up to Month 88
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 4 | 1
nmol/L
  BL: Male Testosterone: number analyzed (Participants) | 3 | 1
  BL: Male Testosterone | 7.53 (4.076) | 7.10 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 22: Male Testosterone | 6.55 (4.751) | 2.40 (NA) — NA: SD could not be calculated as there was only 1 patient.
  WK 70: Male Testosterone: number analyzed (Participants) | 3 | 1
  WK 70: Male Testosterone | 5.17 (1.504) | 32.60 (NA) — NA: SD could not be calculated as there was only 1 patient.
  LOV: Male Testosterone | 8.15 (7.859) | 0.00 (NA) — NA: SD could not be calculated as there was only 1 patient.

15. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Fasting Glucose
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
mg/dL
  BL | 108.1 (55.12) | 96.3 (14.43)
  WK 22: number analyzed (Participants) | 13 | 4
  WK 22 | -14.5 (32.45) | -16.3 (14.93)
  WK 70: number analyzed (Participants) | 10 | 4
  WK 70 | -22.5 (36.87) | -20.8 (24.62)
  LOV | -17.9 (35.99) | -13.8 (22.88)

16. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Hemoglobin A1C (HbA1C) (Glycosylated Hemoglobin)
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Part II Core: Follow-up Cohort: Participants took an ascending dose from 2mg bid or 5 mg bid, up to 30 mg bid and participated in the Part ll Core Follow-up of this study. These patients were patients who transferred from Part l Core phase of the study.
Arm/Group | Part II Core: Expansion Cohort | Part II Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
Percentage
  BL: number analyzed (Participants) | 13 | 4
  BL | 5.7 (0.77) | 6.0 (0.61)
  WK 22: number analyzed (Participants) | 11 | 4
  WK 22 | -0.1 (0.27) | -0.3 (0.28)
  WK 70: number analyzed (Participants) | 8 | 4
  WK 70 | -0.1 (0.43) | -0.6 (0.74)
  LOV: number analyzed (Participants) | 11 | 4
  LOV | -0.1 (0.56) | -0.4 (0.49)

17. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Cholesterol, LDL Cholesterol, HDL Cholesterol, Triglycerides
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmo1/L
Groups:
- Part ll Core: Expansion Cohort: Participants took an ascending dose from 2mg bid or 5 mg bid, up to 30 mg bid and participated in the Part ll Core Expansion of this study. These patients were all newly enrolled into the phase ll part of the study.
Arm/Group | Part ll Core: Expansion Cohort | Part II Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
mmo1/L
  BL Cholesterol | 5.2 (1.36) | 5.7 (1.44)
  WK 22 Cholesterol: number analyzed (Participants) | 13 | 4
  WK 22 Cholesterol | -0.7 (1.58) | -0.5 (0.56)
  WK 70 Cholesterol: number analyzed (Participants) | 10 | 4
  WK 70 Cholesterol | -0.1 (1.35) | -1.2 (1.74)
  LOV Cholesterol | 0.5 (2.39) | 1.5 (5.22)
  BL LDL Cholesterol | 3.0 (1.32) | 4.8 (2.31)
  WK 22 LDL Cholesterol: number analyzed (Participants) | 13 | 4
  WK 22 LDL Cholesterol | -0.3 (1.35) | -1.5 (1.98)
  WK 70 LDL Cholesterol: number analyzed (Participants) | 10 | 4
  WK 70 LDL Cholesterol | 0.0 (1.17) | -2.2 (2.11)
  LOV LDL Cholesterol | 0.3 (1.58) | -0.7 (1.83)
  BL HDL Cholesterol | 1.6 (0.39) | 2.1 (1.85)
  WK 22 HDL Cholesterol: number analyzed (Participants) | 13 | 4
  WK 22 HDL Cholesterol | -0.3 (0.32) | -0.9 (1.58)
  WK 70 HDL Cholesterol: number analyzed (Participants) | 10 | 4
  WK 70 HDL Cholesterol | -0.3 (0.42) | -0.9 (1.60)
  LOV HDL Cholesterol | 0.1 (0.66) | -0.0 (0.49)
  BL Triglycerides | 1.5 (0.70) | 1.4 (0.32)
  WK 22 Triglycerides: number analyzed (Participants) | 13 | 4
  WK 22 Triglycerides | -0.1 (0.42) | 0.1 (0.49)
  WK 70 Triglycerides: number analyzed (Participants) | 10 | 4
  WK 70 Triglycerides | 0.3 (0.76) | -0.2 (0.25)
  LOV Triglycerides | 0.1 (0.64) | -0.1 (0.54)

18. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Sitting Diastolic Blood Pressure (DBP), Sitting Systolic Blood Pressure (SBP)
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Part ll Core: Expansion Cohort | Part II Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
mmHG
  BL DBP | 84.5 (7.01) | 87.3 (4.21)
  WK 22 DPB: number analyzed (Participants) | 13 | 3
  WK 22 DPB | 0.8 (9.59) | 2.6 (11.36)
  WK 70 DPB: number analyzed (Participants) | 10 | 4
  WK 70 DPB | -3.4 (11.65) | -5.8 (12.14)
  LOV DPB | -1.3 (9.23) | -3.2 (7.07)
  BL SBP | 133.2 (12.51) | 130.3 (7.75)
  WK 22 SPB: number analyzed (Participants) | 13 | 4
  WK 22 SPB | -4.0 (12.46) | 8.8 (24.74)
  WK 70 SPB: number analyzed (Participants) | 10 | 4
  WK 70 SPB | -9.5 (15.78) | -4.7 (26.09)
  LOV SPB | -6.2 (16.50) | 0.3 (20.60)

19. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Weight
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Part ll Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
Kg
  BL | 85.4 (23.52) | 84.0 (23.32)
  WK 22: number analyzed (Participants) | 13 | 4
  WK 22 | -2.1 (4.02) | 0.6 (2.64)
  WK 70: number analyzed (Participants) | 10 | 4
  WK 70 | -5.2 (4.56) | -3.2 (5.61)
  LOV | -4.5 (6.68) | -4.4 (7.00)

20. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Body Mass Index (BMI)
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Part ll Core: Expansion Cohort | Part II Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
Kg/m^2
  BL | 30.6 (7.46) | 31.3 (5.49)
  WK 22: number analyzed (Participants) | 13 | 4
  WK 22 | -0.7 (1.42) | 0.2 (1.09)
  WK 70: number analyzed (Participants) | 10 | 4
  WK 70 | -1.9 (1.93) | -1.4 (2.25)
  LOV | -1.6 (2.73) | -2.0 (2.73)

21. Secondary Outcome: Actual Change From BL in Cardiovascular and Other Metabolic Parameters: Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: Improving metabolic abnormalities was assessed by descriptive statistics on the change from baseline. QUICKI is the quantitative insulin sensitivity check index and is derived using the inverse of the sum of algorithms (base 10) of the fasting insulin and fasting glucose: 1/(log(fasting insulin mU/mL)+log(fasting glucose mg/dL)).
  Values typically associated with the QUICKI calculation for insulin resistance in humans fall broadly within a range between 0.45 for unusually healthy individuals and 0.30 in diabetics. So lower numbers reflect greater insulin resistance.
Time Frame: Baseline, Week 22, Week 70, Last observed value, up to Month 88
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Part ll Core: Expansion Cohort | Part II Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
unitless
  BL: number analyzed (Participants) | 13 | 4
  BL | 0.3 (0.03) | 0.3 (0.02)
  WK 22: number analyzed (Participants) | 11 | 4
  WK 22 | 0.0 (0.02) | 0.0 (0.01)
  WK 70: number analyzed (Participants) | 8 | 4
  WK 70 | 0.0 (0.03) | 0.0 (0.06)
  LOV: number analyzed (Participants) | 13 | 4
  LOV | 0.0 (0.04) | 0.0 (0.04)

22. Secondary Outcome: Pharmacokinetics (PK) Parameters: Area Under Curve (AUC)0-6h ss, AUC0-12h ss
Description: Trough PK concentrations and PK profiles at steady-state were collected. The AUC from time 0 to 12 h post dose at steady state, calculated by using the predose concentration (Ctrough,ss) as the 12 h concentration, assuming steady-state has been reached.
Time Frame: pre-dose (0 hour), 1, 1.5, 2, 4 and 6 hours post AM dose for escalation dose or pre-dose (trough) for maintained dose
Population: Pharmacokinetic Analysis Set (PAS): all enrolled patients with at least 1 dose of study drug and at least 1 post-dose PK assessment after Protocol Amendment 4 or after re-entering the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr•ng/mL
Groups:
- 2mg Bid: Participants in the Expansion cohort who took 2mg of osilodrostat
- 5mg Bid: Participants in the Expansion cohort who took 5mg of osilodrostat
- 10mg Bid: Participants in the Expansion cohort who took 10mg of osilodrostat
- 20mg Bid: Participants in the Expansion cohort who took 20mg of osilodrostat
- 30mg Bid: Participants in the Expansion cohort who took 30mg of osilodrostat
Arm/Group | 2mg Bid | 5mg Bid | 10mg Bid | 20mg Bid | 30mg Bid
Number analyzed (Participants) | 4 | 13 | 6 | 1 | 1
hr•ng/mL
  AUC0-6h,ss | 37.79 (42.7) | 94.21 (37.0) | 236.83 (29.9) | NA (NA) — NA: geo-mean/coefficient variation (CV) geo-mean could not be calculated as only 1 patient | NA (NA) — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient
  AUC0-12h,ss: number analyzed (Participants) | 3 | 13 | 6 | 1 | 1
  AUC0-12h,ss | 69.96 (32.6) | 140.65 (43.9) | 339.62 (37.6) | NA (NA) — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient | NA (NA) — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient

23. Secondary Outcome: PK Parameters: Cmax ss, Ctrough ss
Description: Trough PK concentrations and PK profiles at steady-state were collected.
Time Frame: pre-dose (0 hour), 1, 1.5, 2, 4 and 6 hours post AM dose for escalation dose or pre-dose (trough) for maintained dose
Population: PAS: all enrolled patients with at least 1 dose of study drug and at least 1 post-dose PK assessment after Protocol Amendment 4 or after re-entering the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 2mg Bid | 5mg Bid | 10mg Bid | 20mg Bid | 30mg Bid
Number analyzed (Participants) | 6 | 14 | 8 | 2 | 1
ng/mL
  Cmax,ss: number analyzed (Participants) | 4 | 13 | 6 | 1 | 1
  Cmax,ss | 8.76 (46.1) | 23.09 (31.5) | 59.17 (25.5) | NA (NA) — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient | NA (NA) — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient
  Ctrough, ss | 2.73 (49.1) | 4.30 (112.9) | 10.60 (104.8) | 19.69 (53.6) | NA (NA) — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient

24. Secondary Outcome: PK Parameters: Tmax ss,
Description: Trough PK concentrations and PK profiles at steady-state were collected.
Time Frame: pre-dose (0 hour), 1, 1.5, 2, 4 and 6 hours post AM dose for escalation dose or pre-dose (trough) for maintained dose
Population: as for outcome 23
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | 2mg Bid | 5mg Bid | 10mg Bid | 20mg Bid | 30mg Bid
Number analyzed (Participants) | 4 | 13 | 6 | 1 | 1
hour (hr) | 1.50 [1.0 to 4.1] | 1.50 [1.0 to 4.0] | 1.26 [1.0 to 2.0] | NA [NA to NA] — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient | NA [NA to NA] — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient

25. Secondary Outcome: PK Parameters: T1/2 ss,
Description: Trough PK concentrations and PK profiles at steady-state were collected.
Time Frame: pre-dose (0 hour), 1, 1.5, 2, 4 and 6 hours post AM dose for escalation dose or pre-dose (trough) for maintained dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Arm/Group | 2mg Bid | 5mg Bid | 10mg Bid | 20mg Bid | 30mg Bid
Number analyzed (Participants) | 2 | 11 | 6 | 1 | 1
hour (hr) | 6.39 (13.8) | 3.54 (49.8) | 4.32 (47.8) | NA — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient | NA — NA: geo-mean/CV geo-mean could not be calculated as only 1 patient

26. Secondary Outcome: Percentage of Participants Who Were Responders on 24-hour Urine Free Cortisol (UFC) at Week 22
Description: A patient was considered to be a responder if his/her mean UFC level from the three 24-hour urine samples collected at Week 22 was ≤ ULN (as defined by the local laboratories) or represented a ≥50% decrease from baseline. Participants with controlled or partially controlled UFC were defined as: Controlled UFC: mean UFC level <= upper limit of normal (ULN).
  Partially controlled UFC: mean UFC level > ULN but with >= 50% reduction from baseline.
Time Frame: Week 22
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage pf participants
Arm/Group | Part II Core: Expansion Cohort | Part ll Core: Follow-up Cohort
Number analyzed (Participants) | 15 | 4
Percentage pf participants
  Responders | 80.0 [51.91 to 95.67] | 75.0 [19.41 to 99.37]
  Controlled UFC responders | 80.0 [51.91 to 95.67] | 75.0 [19.41 to 99.37]
  Partially controlled UFC responders | 0 [0.00 to 21.80] | 0 [0.00 to 60.24]

27. Secondary Outcome: Number of Participants With Escape
Description: Escape is defined as loss of UFC control (i.e. UFC > ULN) on at least 2 consecutive visits at the highest tolerated dose after previously attaining UFC normalization)
Time Frame: approx. 7 years
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Part l: Core Cohort | Part II Core: Expansion Cohort
Number analyzed (Participants) | 15 | 4
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected from first dose of study treatment until end of study treatment plus 28 days post treatment, up to maximum duration of 350.6 weeks.
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment plus the 28 days post treatment
Arm/Group | Part l: Core Cohort | Part ll Core: Expansion Cohort | Part ll Core: Follow-up Cohort
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/12 | 5/15 | 1/4
Other Adverse Events (participants affected / at risk) | 12/12 | 15/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part l: Core Cohort (N=12) | Part ll Core: Expansion Cohort (N=15) | Part ll Core: Follow-up Cohort (N=4)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Takayasu's arteritis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part l: Core Cohort (N=12) | Part ll Core: Expansion Cohort (N=15) | Part ll Core: Follow-up Cohort (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 6 | 2
Diabetes insipidus (Endocrine disorders) | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 | 2 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 8 | 2
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2
Asthenia (General disorders) | 0 | 5 | 2
Chest discomfort (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 3 | 3
Feeling drunk (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 1 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 0 | 4 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 3 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 1
Furuncle (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 2
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Tongue fungal infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 3
Viral rhinitis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 2
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aldosterone urine increased (Investigations) | 0 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Blood aldosterone decreased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood corticotrophin increased (Investigations) | 0 | 5 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 4 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood gonadotrophin abnormal (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood luteinising hormone decreased (Investigations) | 0 | 1 | 0
Blood phosphorus (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0
Blood prolactin increased (Investigations) | 0 | 0 | 1
Blood testosterone free increased (Investigations) | 0 | 0 | 1
Blood testosterone increased (Investigations) | 0 | 2 | 4
Blood uric acid increased (Investigations) | 1 | 1 | 0
Cortisol decreased (Investigations) | 0 | 0 | 1
Cortisol free urine decreased (Investigations) | 0 | 0 | 1
Cortisol free urine increased (Investigations) | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Gastric pH decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 1 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0
Hormone level abnormal (Investigations) | 0 | 4 | 3
Lipase increased (Investigations) | 2 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 2
Oestradiol increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Protein total increased (Investigations) | 0 | 1 | 0
Renin decreased (Investigations) | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0
Urine leukocyte esterase (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 2 | 0
Weight increased (Investigations) | 1 | 2 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyposideraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cold-stimulus headache (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 6 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Abnormal sleep-related event (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Melanoderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 3 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT01331239/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT01331239/SAP_001.pdf